CLINICAL TRIAL: NCT06955286
Title: Study on the Incidence of Adrenal Insufficiency After Surgery in Primary Aldosteronism Patients Concurrent With or Without Autonomous Cortisol Secretion
Status: Recruiting | Type: Observational
Sponsor: Qifu Li (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: 2025-040-01
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Primary Aldosteronism; Autonomous Cortisol Secretion; Adrenal Insufficiency
Keywords: Primary Aldosteronism; Autonomous Cortisol Secretion; Adrenal Insufficiency; ACTH stimulation test
MeSH Terms: conditions — Hyperaldosteronism; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients With Primary Aldosteronism Concurrent With or Without Autonomous Cortisol Secretion: primary aldosteronism patients concurrent with autonomous cortisol secretion underwent surgical treatment and completed the ACTH stimulation test
  Interventions: Diagnostic Test: complete ACTH stimulation test the day after surgery

INTERVENTIONS:
Diagnostic Test: complete ACTH stimulation test the day after surgery — patients complete ACTH stimulation test on the one day after surgery

SUMMARY:
To evaluate the incidence of adrenal insufficiency after surgery in Primary aldosteronism (PA) patients concurrent with or without autonomous cortisol secretion (ACS).

DETAILED DESCRIPTION:
This study is a prospective, single-center research. Primary aldosteronism patients concurrent with or without autonomous cortisol secretion who underwent adrenalectomy and completed the adrenocorticotropic hormone (ACTH) stimulation test will be included. To evaluate the incidence of adrenal insufficiency after surgery in these patients.

ELIGIBILITY:
Inclusion Criteria:

* PA conccurent with or without autonomous cortisol secretion
* complete adrenalectomy
* complete ACTH stimulation test on the one day after surgery
* complete follow-up at 6，12 months after surgery

Exclusion Criteria:

* Patients underwent partial adrenalectomy
* Suspicion of familial hyperaldosteronism or Liddle syndrome. [i.e., age <20 years, hypertension and hypokalemia, or with family history]
* Suspicion of pheochromocytoma or adrenal carcinoma.
* Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV; History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 3 months; Severe anemia (Hb<60g/L); Serious liver dysfunction or chronic kidney disease aspartate aminotransferase (AST) or alanine transaminase (ALT) >3 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2); Systemic Inflammatory Response Syndrome (SIRS); Uncontrolled diabetes (FBG≥13.3 mmol/L); Obesity (BMI≥35 kg/m2) or Underweight (BMI≤18 kg/m2); Untreated aneurysm; Other comorbidity potentially interfering with treatment;
* Patients with actively malignant tumor.
* Long- term use of glucocorticoids.
* Suspected PBMAH or PPNAD;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Aldosteronism Patients Concurrent With or Without Autonomous Cortisol Secretion who underwent surgery and completed the ACTH stimulation test
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the Incidence of Adrenal Insufficiency After Surgery | the one day after surgery
  the Incidence of Adrenal Insufficiency After Surgery on the one day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, China, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Libianto R, Russell GM, Stowasser M, Gwini SM, Nuttall P, Shen J, Young MJ, Fuller PJ, Yang J. Detecting primary aldosteronism in Australian primary care: a prospective study. Med J Aust. 2022 May 2;216(8):408-412. doi: 10.5694/mja2.51438. Epub 2022 Feb 25. PMID 35218017
- [Result] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Result] Nakajima Y, Yamada M, Taguchi R, Satoh T, Hashimoto K, Ozawa A, Shibusawa N, Okada S, Monden T, Mori M. Cardiovascular complications of patients with aldosteronism associated with autonomous cortisol secretion. J Clin Endocrinol Metab. 2011 Aug;96(8):2512-8. doi: 10.1210/jc.2010-2743. Epub 2011 May 18. PMID 21593113
- [Result] Naruse M, Katabami T, Shibata H, Sone M, Takahashi K, Tanabe A, Izawa S, Ichijo T, Otsuki M, Omura M, Ogawa Y, Oki Y, Kurihara I, Kobayashi H, Sakamoto R, Satoh F, Takeda Y, Tanaka T, Tamura K, Tsuiki M, Hashimoto S, Hasegawa T, Yoshimoto T, Yoneda T, Yamamoto K, Rakugi H, Wada N, Saiki A, Ohno Y, Haze T. Japan Endocrine Society clinical practice guideline for the diagnosis and management of primary aldosteronism 2021. Endocr J. 2022 Apr 28;69(4):327-359. doi: 10.1507/endocrj.EJ21-0508. Epub 2022 Apr 12. PMID 35418526
- [Result] Araujo-Castro M, Paja Fano M, Pla Peris B, Gonzalez Boillos M, Pascual-Corrales E, Garcia-Cano AM, Parra Ramirez P, Rojas-Marcos PM, Ruiz-Sanchez JG, Vicente A, Gomez-Hoyos E, Ferreira R, Garcia Sanz I, Recasens M, Barahona San Millan R, Picon Cesar MJ, Diaz Guardiola P, Perdomo C, Manjon L, Garcia-Centeno R, Percovich JC, Rebollo Roman A, Gracia Gimeno P, Robles Lazaro C, Morales M, Calatayud M, Collao SAF, Meneses D, Sampedro Nunez MA, Escudero Quesada V, Ribas EM, Sanmartin Sanchez A, Diaz CG, Lamas C, Guerrero-Vazquez R, Del Castillo Tous M, Serrano J, Michalopoulou T, Moya Mateo EM, Hanzu F. Autonomous cortisol secretion in patients with primary aldosteronism: prevalence and implications on cardiometabolic profile and on surgical outcomes. Endocr Connect. 2023 Aug 2;12(9):e230043. doi: 10.1530/EC-23-0043. PMID 37410097
- [Result] Fujimoto K, Honjo S, Tatsuoka H, Hamamoto Y, Kawasaki Y, Matsuoka A, Ikeda H, Wada Y, Sasano H, Koshiyama H. Primary aldosteronism associated with subclinical Cushing syndrome. J Endocrinol Invest. 2013 Sep;36(8):564-7. doi: 10.3275/8818. Epub 2013 Feb 4. PMID 23385627
- [Result] Katabami T, Matsuba R, Kobayashi H, Nakagawa T, Kurihara I, Ichijo T, Tsuiki M, Wada N, Ogawa Y, Sone M, Inagaki N, Yoshimoto T, Takahashi K, Yamamoto K, Izawa S, Kakutani M, Tanabe A, Naruse M. Primary aldosteronism with mild autonomous cortisol secretion increases renal complication risk. Eur J Endocrinol. 2022 Apr 25;186(6):645-655. doi: 10.1530/EJE-21-1131. PMID 35380982
- [Result] Wu WC, Peng KY, Lu JY, Chan CK, Wang CY, Tseng FY, Yang WS, Lin YH, Lin PC, Chen TC, Huang KH, Chueh JS, Wu VC. Cortisol-producing adenoma-related somatic mutations in unilateral primary aldosteronism with concurrent autonomous cortisol secretion: their prevalence and clinical characteristics. Eur J Endocrinol. 2022 Sep 14;187(4):519-530. doi: 10.1530/EJE-22-0286. Print 2022 Oct 1. PMID 35900323
- [Result] Liao YY, Song Y, Hu JB, Yang SM, Zheng Y, Li QF. [Clinical characteristics and prognosis of primary aldosteronism associated with subclinical Cushing syndrome]. Zhonghua Nei Ke Za Zhi. 2024 Apr 1;63(4):378-385. doi: 10.3760/cma.j.cn112138-20230830-00100. Chinese. PMID 38561283
- [Result] DeLozier OM, Dream SY, Findling JW, Carroll TB, Evans DB, Wang TS. Selective Glucocorticoid Replacement Following Unilateral Adrenalectomy for Hypercortisolism and Primary Aldosteronism. J Clin Endocrinol Metab. 2022 Jan 18;107(2):e538-e547. doi: 10.1210/clinem/dgab698. PMID 34558612
- [Result] Gerards J, Heinrich DA, Adolf C, Meisinger C, Rathmann W, Sturm L, Nirschl N, Bidlingmaier M, Beuschlein F, Thorand B, Peters A, Reincke M, Roden M, Quinkler M. Impaired Glucose Metabolism in Primary Aldosteronism Is Associated With Cortisol Cosecretion. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3192-3202. doi: 10.1210/jc.2019-00299. PMID 30865224